CLINICAL TRIAL: NCT01802255
Title: Study of the Safety of Administration of Sevoflurane for Long-term Critically Ill Patients Sedation Undergoing Mechanical Ventilation. Prospective, Controlled, Randomized, Multicenter, Clinical Trial.
Brief Title: Sevoflurane- Safety in Long-term Sedation Procedures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment in the Centres
Sponsor: F Javier Belda (Other)
Responsible Party: Sponsor-Investigator, F Javier Belda, Prof. Dr. F Javier Belda, Fundación para la Investigación del Hospital Clínico de Valencia
Organization: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ECSEVO-LT-011; 2011-002555-34 (EudraCT Number)
Record Dates: First submitted 2013-02-09; First posted 2013-03-01 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Poisoning by Inhaled Anaesthetic; Fluoride Poisoning; Recovery From Sedation; Renal Function; Hepatic Function
Keywords: Inhalatory sedation; Sevoflurane; AnaConDa; Nephrotoxicity; Hepatotoxicity; Midazolam; Propofol
MeSH Terms: conditions — Fluoride Poisoning | interventions — Sevoflurane; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhalatory sedation (Experimental): Sevoflurane given via AnaConDa for sedation minimum 48 hours
  Interventions: Drug: Sevoflurane
- Intravenous sedation (Active Comparator): Midazolam given intravenously for sedation minimum 48 hours
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Sevoflurane — Sedation with inhaled anesthetic via AnaConDa.
  Other Names: Sevorane, Ultane, Sojourn
  Arms: Inhalatory sedation
Drug: Midazolam — Intravenous sedation.
  Other Names: Versed
  Arms: Intravenous sedation

SUMMARY:
Patients needing intensive care often require sedative drugs to reduce anxiety and agitation during ventilator care and invasive therapeutic and diagnostic procedures. At present there is no optimal sedative agent for these patients. The most commonly used sedative agents in intensive care units are midazolam and propofol. Both drugs have side effects of clinical importance.

At present, a viable alternative to intravenous sedation is inhalatory sedation. Sevoflurane, as other inhaled anesthetic agents, is sedative in low doses. A new simplified method of administration of isoflurane or sevoflurane has been developed. The Anesthetic Conserving Device is a modified heat-moisture exchanger (HME) that permits direct infusion of sevoflurane to the airway, where it is vaporized in an evaporator rod in the device.

However, the use of sevoflurane is limited to anesthesia and sedation lasting no more than 12 hours, since the possible renal problems posed by inorganic fluoride in prolonged operations remain the subject of controversy.

The primary aim (and primary hypothesis) of the current trial is to determine whether sevoflurane can be administered as a sedative drug for more than 48 hours without clinically relevant physiopathological effects on kidney and liver function.

Other end-points of the trial are to evaluate the quality of sedation of sevoflurane, in terms of sedation control, the rapidity and predictability of awakening, and the incidence of delirium in critical care patients.

ELIGIBILITY:
Inclusion Criteria:

* Signing of the informed consent document (patient or relatives).
* Patient age 18 years or older.
* Expected minimum duration of sedation: 48 hours.

Exclusion Criteria:

* Chronic renal failure treated with replacement therapy (hemodialysis or peritoneal dialysis).
* Acute kidney injury in Stage 3 of AKIN classification
* Grade C hepatic Child-Pugh classification
* Established Acute Respiratory Distress Syndrome (ARDS).
* Central nervous system pathology with cognitive disorders that not allow performing the test of the study: severe dementia, Alzheimer's disease, depression, schizophrenia, acute stroke.
* Head trauma with Glasgow <12.
* Patient treated with antiepileptic drugs that must be maintained during the study period
* Patients requiring the use of neuromuscular blocking agents during the infusion of study drug, except for the insertion of the endotracheal tube.
* Epidural or spinal analgesia
* Allergy or known hypersensitivity to any of the study drugs
* Patients with known or suspected genetic susceptibility to malignant hyperthermia
* Previous participation in this trial
* Participation in another clinical trial within 4 weeks prior to selection.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Maintenance of renal function. | Baseline. Posteriorly, every 12 hours for the full length of sedation. After sedation, every 24 hours up to one week
  Measurements in plasma: creatinine and cystatin levels.

SECONDARY OUTCOMES:
Assessment of liver function | Baseline. Posteriorly, every 12 hours for the full length of sedation. After sedation, every 24 hours up to one week
  Measurements in plasma: SGOT (aspartate aminotransferase, AST), SGPT (alanine aminotransferase, ALT), LDH (lactate dehydrogenase) alkaline phosphatase, conjugated and total bilirubin, cholesterol, triglycerides, albumin, total proteins, electrolytes and glycogen.
Plasma pharmacokinetics of fluoride | Baseline. Posteriorly, every 12 hours for the full length of sedation. After sedation, every 24 hours up to one week
  Determine evolutionary plasmatic levels of fluorides.
Incidence of delirium | Baseline. Posteriorly, every 12 hours for the full length of sedation. After sedation, every 24 hours up to one week
  The incidence of delirium will be evaluated by the CAM-ICU method.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Soro, MD, PhD, Study Director — Hospital Clínico Universitario de Valencia; Luciano Aguilera, MD, PhD, Principal Investigator — Hospital de Basurto; Carlos Soria, MD, PhD, Principal Investigator — Complejo Asistencial de León; Francisco Acosta, MD, PhD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be anonymous

REFERENCES:
- [Background] Kong KL, Bion JF. Sedating patients undergoing mechanical ventilation in the intensive care unit--winds of change? Br J Anaesth. 2003 Mar;90(3):267-9. doi: 10.1093/bja/aeg066. No abstract available. PMID 12594134
- [Background] Rohm KD, Wolf MW, Schollhorn T, Schellhaass A, Boldt J, Piper SN. Short-term sevoflurane sedation using the Anaesthetic Conserving Device after cardiothoracic surgery. Intensive Care Med. 2008 Sep;34(9):1683-9. doi: 10.1007/s00134-008-1157-x. Epub 2008 May 24. PMID 18500419